CLINICAL TRIAL: NCT02038075
Title: Brief Cognitive Behavioral Therapy for Military Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: University of Memphis (Other); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Craig Bryan, Executive Director, National Center for Veterans Studies, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W81XWH-09-1-0569; W81XWH-09-1-0569 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Suicide; Suicidal Ideation
Keywords: suicide; suicidal ideation; military; veteran; cognitive behavioral therapy; behavioral therapy; psychotherapy; Brief Cognitive Behavioral Therapy (BCBT); Treatement As Usual (TAU)
MeSH Terms: conditions — Suicide; Suicidal Ideation | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Cognitive Behavioral Therapy (BCBT) (Experimental): In addition to TAU, participants in BCBT receive 12 outpatient individual psychotherapy sessions scheduled on a weekly or biweekly basis, with the first session lasting 90 minutes and subsequent sessions lasting 60 minutes. BCBT was is delivered in three sequential phases. In phase I (5 sessions), the therapist identifies patient-specific factors that contribute to and maintain suicidal behaviors, provides a cognitive-behavioral conceptualization, collaboratively develops a crisis response plan, and teaches basic emotion regulation skills. In phase II (5 sessions), the therapist applies cognitive strategies to reduce beliefs and assumptions that serve as vulnerabilities to suicidal behavior. In phase III (2 sessions), a relapse prevention task is conducted.
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy (BCBT)
- Treatment As Usual (TAU) (Active Comparator): Participants in TAU receive usual care from military clinicians as well as non-military clinicians from the local community, as determined by participants' primary mental health care provider. All mental health, substance abuse, and medical treatment are provided within the military health care system at no cost to participants.
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy (BCBT)
  Other Names: Cognitive Therapy
  Arms: Brief Cognitive Behavioral Therapy (BCBT)
Behavioral: Treatment As Usual (TAU)
  Other Names: Usual Care; Enhanced Treatment As Usual; Enhanced Care; Enhanced Care As Usual
  Arms: Treatment As Usual (TAU)

SUMMARY:
The primary purpose of this study is to compare the effectiveness of brief cognitive-behavioral therapy (B-CBT) for the treatment of suicidality, including suicidal ideation and attempts (regardless of Axis I or II diagnosis) among active duty military personnel. The standard null hypothesis will involve tests conducted comparing improvement following B-CBT (treatment duration of 12 weeks) to treatment as usual (TAU). The primary outcome comparisons will include both direct markers of suicidality (i.e. suicide, suicide attempts) and indirect markers including associated symptomatology (i.e. suicidal ideation, intent, anxiety, depression, hopelessness, substance abuse, and sleep disturbance), along with remission of psychiatric diagnoses. Secondary purposes include the prospective investigation of suicide risk factors and warning signs to explore these variables' ability to predict subsequent suicidal behavior following an index attempt.

DETAILED DESCRIPTION:
The research gap in the treatment of suicidality is considerable, particularly with military populations, including those returning from deployment in support of OIF/OEF. Only one randomized clinical trial targeting suicidality has been conducted with a military sample (Rudd et al., 1996). Although time-limited treatment of suicidality is the primary target of the project, additional elements will be explored including prospective investigation of suicide risk factors and warning signs, as well as development of a centralized software assessment/management tracking system for high-risk suicidal individuals. Reference to "active duty" refers to U.S. military service members that have been activated and deployed as a part of OIF/OEF in accordance with federal orders under Title 10 or 32, Unites States Code. This includes individuals on active duty from the National Guard and Reserve forces.

Specific Aim 1: To evaluate the effectiveness of brief cognitive-behavioral therapy (B-CBT) for the treatment of suicidality, including suicidal ideation and attempts (regardless of Axis I or II diagnosis) among active duty military personnel. It is anticipated that a large percentage of those identified for treatment will include military personnel recently returned from OIF/OEF. The standard null hypothesis will involve tests conducted comparing improvement following B-CBT (treatment duration of 12 weeks) to treatment as usual (TAU). The primary outcome comparisons will include both direct markers of suicidality (i.e. suicide, suicide attempts) and indirect markers including associated symptomatology (i.e. suicidal ideation, intent, anxiety, depression, hopelessness, substance abuse, agitation, and sleep disturbance), along with remission of psychiatric diagnoses.

Specific Aim 2: To engage in prospective investigation of suicide risk factors (i.e. psychiatric diagnosis and history, suicidal ideation, intent, anxiety, depression, hopelessness) and warning signs (i.e. agitation, sleep disturbance), exploring their ability to predict subsequent suicidal behavior following onset of suicidality.

Specific Aim 3: To explore the effectiveness of B-CBT (versus TAU) for increasing appropriate utilization of and compliance with medical, mental health, and substance abuse treatment, as well as improving psychological and social functioning.

Specific Aim 4: To develop a risk management software program for the initial risk assessment, ongoing monitoring and clinical management of high-risk suicidal patients. The software program would provide a mechanism for organizing and tracking clinical risk factors and warning signs for suicide, along with appropriate management and clinical intervention strategies during the treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military
* 18 years or older
* Current suicidal ideation with intent to die and/or suicide attempt within past month
* Able to complete informed consent procedures

Exclusion Criteria:

* Psychiatric or medical condition that precludes informed consent or outpatient therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2011-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Rudd, PhD, ABPP, Principal Investigator — National Center for Veterans Studies & The University of Utah; Craig J Bryan, PsyD, ABPP, Study Director — National Center for Veterans Studies & The University of Utah
Locations (1):
- Fort Carson, Colorado Springs, Colorado, United States

REFERENCES:
- [Background] Bryan CJ, Rudd MD, Wertenberger E. Reasons for suicide attempts in a clinical sample of active duty soldiers. J Affect Disord. 2013 Jan 10;144(1-2):148-52. doi: 10.1016/j.jad.2012.06.030. Epub 2012 Aug 1. PMID 22858207
- [Background] Bryan CJ, Rudd MD. Life stressors, emotional distress, and trauma-related thoughts occurring in the 24 h preceding active duty U.S. soldiers' suicide attempts. J Psychiatr Res. 2012 Jul;46(7):843-8. doi: 10.1016/j.jpsychires.2012.03.012. Epub 2012 Apr 1. PMID 22464944
- [Result] Rudd MD, Bryan CJ, Wertenberger EG, Peterson AL, Young-McCaughan S, Mintz J, Williams SR, Arne KA, Breitbach J, Delano K, Wilkinson E, Bruce TO. Brief cognitive-behavioral therapy effects on post-treatment suicide attempts in a military sample: results of a randomized clinical trial with 2-year follow-up. Am J Psychiatry. 2015 May;172(5):441-9. doi: 10.1176/appi.ajp.2014.14070843. Epub 2015 Feb 13. PMID 25677353
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- See also: National Center for Veterans Studies — http://veterans.utah.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were identified during weekly behavioral health treatment team meetings and daily emergency department reports. All soldiers admitted to inpatient psychiatric hospitalization for suicidal ideation or for a suicide attempt from January 2011 to September 2012 were referred upon discharge for determination of eligibility.
Pre-assignment Details: 30 of 206 referred Soldiers were excluded (15 due to planned move in next 6 months, 15 refused). 24 of 176 consenting to participate were excluded (22 ineligible, 2 dropped before randomization).
Groups:
- Brief Cognitive Behavioral Therapy (BCBT): In addition to TAU, participants in BCBT receive 12 outpatient individual psychotherapy sessions scheduled on a weekly or biweekly basis, with the first session lasting 90 minutes and subsequent sessions lasting 60 minutes. BCBT was is delivered in three sequential phases. In phase I (5 sessions), the therapist identifies patient-specific factors that contribute to and maintain suicidal behaviors, provides a cognitive-behavioral conceptualization, collaboratively develops a crisis response plan, and teaches basic emotion regulation skills. In phase II (5 sessions), the therapist applies cognitive strategies to reduce beliefs and assumptions that serve as vulnerabilities to suicidal behavior. In phase III (2 sessions), a relapse prevention task is conducted.
  Brief Cognitive Behavioral Therapy (BCBT)
- Treatment As Usual (TAU): Participants in TAU receive usual care from military clinicians as well as non-military clinicians from the local community, as determined by participants' primary mental health care provider. All mental health, substance abuse, and medical treatment are provided within the military health care system at no cost to participants.
  Treatment As Usual (TAU)
Period: Overall Study
Arm/Group | Brief Cognitive Behavioral Therapy (BCBT) | Treatment As Usual (TAU)
Started | 76 | 76
Completed | 73 | 76
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Cognitive Behavioral Therapy (BCBT) | Treatment As Usual (TAU) | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.18 (6.25) | 27.62 (621) | 27.40 (6.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 64 | 69 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 21 | 34
  Not Hispanic or Latino | 63 | 55 | 118
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants] — Participants allowed to select more than one racial identity
  participants
    American Indian or Alaska Native | 4 | 3 | 7
    Asian | 1 | 2 | 3
    Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
    Black or African American | 10 | 10 | 20
    White | 58 | 52 | 110
    More than one race | 5 | 7 | 12
    Unknown or Not Reported | 0 | 1 | 1
Military rank [Number; unit: participants]
  E1-E4 | 60 | 51 | 111
  E5-E6 | 15 | 20 | 35
  E7-E9 | 1 | 4 | 5
  Warrant Officer | 0 | 1 | 1
Deployment history [Number; unit: participants]
  None | 18 | 10 | 28
  One | 28 | 31 | 59
  Multiple (2+) | 30 | 35 | 65
Prior suicide attempts [Number; unit: participants]
  None | 17 | 19 | 36
  One | 24 | 34 | 58
  Multiple (2+) | 35 | 23 | 58
Psychiatric diagnosis (SCID) [Number; unit: participants] — Only includes diagnoses occurring in 5% or greater of participants in at least one treatment arm. Determined using Structured Clinical Interview for DSM-IV, Axis I and Axis II.
  participants
    Major depressive | 55 | 63 | 118
    Posttraumatic stress | 26 | 34 | 60
    Substance dependence | 13 | 7 | 20
    Alcohol dependence | 11 | 7 | 18
    Social phobia | 7 | 5 | 12
    Panic | 4 | 3 | 7
    Anxiety | 4 | 2 | 6
    Depressive personality | 9 | 5 | 14
    Borderline personality | 7 | 8 | 15
    Antisocial personality | 5 | 3 | 8
Medications [Number; unit: participants] — Based on self-report and medical record review
  participants
    Antidepressant | 47 | 47 | 94
    Anticonvulsant | 9 | 5 | 14
    Antihypertensive | 11 | 16 | 27
    Antipsychotic | 10 | 13 | 23
    Anxiolytic | 3 | 2 | 5
    Benzodiazepine | 6 | 12 | 18
    Muscle relaxer | 6 | 2 | 8
    Opioid | 6 | 7 | 13
    Opioid antagonis | 3 | 1 | 4
    Sleep/hypnotic | 12 | 14 | 26
    Stimulant | 2 | 3 | 5
    Other | 16 | 18 | 34
Beck Scale for Suicide Ideation, Current [Mean (Standard Deviation); unit: units on a scale] — The intensity of current (i.e., past week) suicidal ideation was measured using the 19-item self-report Beck Scale for Suicide Ideation. Scores range from 0 to 38, with higher scores indicating more severe thoughts and plans about suicide.
  units on a scale | 10.83 (8.67) | 11.07 (8.43) | 10.95 (8.53)
Beck Scale for Suicide Ideation, Worst [Mean (Standard Deviation); unit: units on a scale] — The intensity of the most severe suicidal ideation since the last assessment period was measured using the 19-item self-report Beck Scale for Suicide Ideation, Worst. Scores range from 0 to 38, with higher scores indicating more severe thoughts and plans about suicide.
  units on a scale | 19.16 (9.30) | 19.07 (8.69) | 19.11 (8.97)
Beck Hopelessness Scale [Mean (Standard Deviation); unit: units on a scale] — The intensity of hopelessness was measured using the 20-item self-report Beck Hopelessness Scale. Scores range from 0 to 20, with higher scores indicating more severe hopelessness.
  units on a scale | 12.87 (6.12) | 12.72 (6.02) | 12.80 (6.05)
Beck Depression Inventory, 2nd Edition [Mean (Standard Deviation); unit: units on a scale] — The intensity of depression symptoms was measured using the 21-item self-report Beck Depression Inventory, Second Edition. Scores range from 0 to 63, with higher scores indicating more severe depression.
  units on a scale | 31.95 (14.26) | 33.51 (13.39) | 32.73 (13.81)
Beck Anxiety Inventory [Mean (Standard Deviation); unit: units on a scale] — The intensity of physiological anxiety symptoms was measured using the 20-item self-report Beck Anxiety Inventory. Scores range from 0 to 60, with higher scores indicating more severe anxiety.
  units on a scale | 28.87 (14.78) | 29.74 (13.96) | 29.30 (14.33)
PTSD Checklist, Military Version [Mean (Standard Deviation); unit: units on a scale] — The intensity of posttraumatic stress symptoms during the past month was measured using the 17-item self-report PTSD Checklist, Military Version. Scores range from 17 to 85, with higher scores indicating more severe PTSD symptoms.
  units on a scale | 55.15 (18.10) | 57.39 (15.63) | 56.27 (16.89)

OUTCOME MEASURES:

1. Primary Outcome: Estimated Percentage of Participants Making Suicide Attempt During 24-month Follow-up
Description: The SASII is a clinician-administered interview designed to assess the factors involved in nonfatal suicide attempts and intentional self-injury. The SASII assesses variables related to method, reliability, lethality, impulsivity, likelihood of rescue, suicidal intent, consequences, and habitual self-injury. Interrater reliabilities for each item range from .87-.98, with the correlation for rater classification of behavior (i.e., suicide attempt or non-suicidal self-injury) being .92. The SASII demonstrates very high agreement in identifying and classifying suicide-related events when compared to clinician therapy notes, patient diary cards, and medical records (for events requiring medical attention).
Time Frame: 24 months
Population: intent to treat
Measure: Number; unit: estimated percentage w/ suicide attempt
Arm/Group | Brief Cognitive Behavioral Therapy (BCBT) | Treatment As Usual (TAU)
Number analyzed (Participants) | 76 | 76
estimated percentage w/ suicide attempt | 13.8 | 40.2
Statistical Analysis 1: Comparison: Brief Cognitive Behavioral Therapy (BCBT) vs Treatment As Usual (TAU); To determine the effectiveness of brief CBT compared with treatment as usual, univariate and multivariate Cox proportional hazard regression models were used to analyze time to the first suicide attempt. Time to suicide attempt was measured by calculating the total number of days from enrollment to the first suicide attempt. For participants without a suicide attempt, the total number of days from enrollment to the last assessment was calculated; Test type: Superiority or Other; p = .02, Regression, Cox; Cox Proportional Hazard = .38, 95% CI 2-sided [.16 to .87]

2. Secondary Outcome: Scale for Suicide Ideation (SSI)
Description: The SSI is a 21-item, interviewer-administered scale used to evaluate the current intensity of the patient's specific attitudes, behaviors, and plans to commit suicide. The SSI has moderately high internal consistency and good concurrent and discriminant validity for psychiatric outpatients. Inter-rater reliability has been found to be higher than .98, with good evidence of predictive validity.
Time Frame: 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Beck Depression Inventory, Second Edition (BDI-II)
Description: The BDI-II is a 21-item self-report instrument developed to measure severity of depression in adults and adolescents. Each of the items consists of four statements reflecting increasing levels of severity for a particular symptom of depression.
Time Frame: 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Beck Hopelessness Scale (BHS)
Description: The BHS consists of 20 true-false statements designed to assess the extent of positive and negative beliefs about the future.
Time Frame: 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Beck Anxiety Inventory
Description: The BAI is a 21-item scale that measures the severity of anxiety in adults and adolescents.
Time Frame: 24 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Structured Clinical Interview for DSM-IV, Axis I and II (SCID)
Description: The SCID (patient version with psychotic screen) is a diagnostic instrument based on DSM-IV diagnostic criteria for Axis I disorders.
Time Frame: Intake
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Suicide Intent Scale
Description: The SIS is a 15-item, interviewer-administered assessment of the intensity of an individual's intent to die at the time of a suicide attempt. It assesses verbal and nonverbal indicators of suicidal attempt including objective circumstances surrounding the attempt, and the attempters' perceptions of the attempt.
Time Frame: 24 months
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Interpersonal Needs Questionnaire (INQ)
Description: The INQ is a 10-item self-report questionnaire that measures current beliefs about the extent to which the respondent feels connected to others (i.e., thwarted belongingness), and the extent to which he or she feels like a burden on the people in their lives (i.e., perceived burdensomeness).
Time Frame: 24 months
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Suicide Cognitions Scale (SCS)
Description: The SCS-R is an 18-item self-report measure that measures two aspects of suicide-specific hopelessness: 1) unlovability (which measures more trait-like aspects of hopelessness), and 2) unbearability (which measures more state-like aspects of hopelessness).
Time Frame: 24 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Post Treatment Health Interview (PTHI)
Description: Frequency, intensity, and location of each patient's accessing of medical services will be assessed via medical record review.
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Brief Cognitive Behavioral Therapy (BCBT) | Treatment As Usual (TAU)
Serious Adverse Events (participants affected / at risk) | 1/76 | 1/76
Other Adverse Events (participants affected / at risk) | 0/76 | 0/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brief Cognitive Behavioral Therapy (BCBT) (N=76) | Treatment As Usual (TAU) (N=76)
Suicide death (Psychiatric disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No